CLINICAL TRIAL: NCT00115245
Title: A Randomized, Open-Label Trial of Telbivudine Versus Adefovir Dipivoxil in Adults With HBegAg-Positive, Compensated Chronic Hepatitis B
Brief Title: Telbivudine Versus Adefovir Dipivoxil in Adults With HBegAg-Positive, Compensated Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV-02B-018
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; adefovir dipivoxil

INTERVENTIONS:
Drug: Telbivudine (LdT)
Drug: Adefovir Dipivoxil

SUMMARY:
This research study is being conducted to compare the safety and effectiveness of the investigational medication, LdT (telbivudine) versus adefovir dipivoxil, a drug approved by the Food and Drug Administration (FDA) for the treatment of hepatitis B infection. The results for patients taking LdT will be compared to results for patients taking adefovir dipivoxil.

ELIGIBILITY:
Inclusion Criteria:

* Documented compensated chronic hepatitis B defined by clinical history compatible with compensated chronic hepatitis B
* Detectable serum HBsAg at the Screening visit

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient is coinfected with hepatitis C virus (HCV), hepatitis D virus (HDV) or HIV
* Patient previously received lamivudine, adefovir dipivoxil, or an investigational anti-hepatitis B virus (HBV) nucleoside or nucleotide analog at any time
* Patient has received interferon or other immunomodulatory treatment for HBV infection in the 12 months before screening for this study

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (4):
  - Los Angeles, California
  - Pasadena, California
  - San Francisco, California
  - Miami, Florida
- Australia (2):
  - Clayton
  - Wooloongabba
- Canada (3):
  - Calgary
  - Toronto
  - Winnipeg
- Hong Kong, China
- Paris, France
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan
- Bangkok, Thailand

REFERENCES:
- [Derived] Chan HL, Heathcote EJ, Marcellin P, Lai CL, Cho M, Moon YM, Chao YC, Myers RP, Minuk GY, Jeffers L, Sievert W, Bzowej N, Harb G, Kaiser R, Qiao XJ, Brown NA; 018 Study Group. Treatment of hepatitis B e antigen positive chronic hepatitis with telbivudine or adefovir: a randomized trial. Ann Intern Med. 2007 Dec 4;147(11):745-54. doi: 10.7326/0003-4819-147-11-200712040-00183. Epub 2007 Oct 1. PMID 17909201